CLINICAL TRIAL: NCT02761239
Title: Descriptive In Vivo Study of Evaluating the Innervation of The Human Cricopharyngeal Muscle By The Recurrent Laryngeal Nerve and External Branch of The Superior Laryngeal Nerve
Brief Title: Innervation of Human Cricopharyngeal Muscle By Recurrent Laryngeal and External Branch of Superior Laryngeal Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Uludag, Associated Professor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SEEAH02
Record Dates: First submitted 2015-09-09; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Larynx
Keywords: cricopharyngeal muscle; innervation by EBSLN; A prospective case-controlled study
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cricopharyngeal muscle innervation (Other): The recurrent laryngeal nerve (RLN), vagus nerve, external branch of the superior laryngeal nerve (EBSLN) and pharyngeal plexus were stimulated intraoperatively by the NIM 3.0 Nerve Monitoring System (Medtronic Xomed, Jacksonville, FL, USA). Responses were evaluated by visual observation of the cricopharyngeal muscle and electromyographies via needle electrodes inserted into the cricopharyngeal muscle.
  Interventions: Device: The NIM 3.0 Nerve Monitoring System

INTERVENTIONS:
Device: The NIM 3.0 Nerve Monitoring System — Electromyography recordings were accomplished with a pair of needle electrodes inserted through the CP muscle, which were plugged into the third and fourth channels of interface-connector box.The recurrent laryngeal nerve(RLN), vagus nerve, external branch of the superior laryngeal nerve(EBSLN) and pharyngeal plexus were stimulated with a current of 1 mA and a frequency of 4 MHz and the event threshold at 100 microV.

SUMMARY:
The investigators hypothesized that, external branch of the superior laryngeal nerve (EBSLN) and/or recurrent laryngeal nerve (RLN) contribute to the motor function of the human cricopharyngeal muscle (CP). The investigators aimed to assess the contribution of the laryngeal nerves (EBSLN and RLN) to the motor activity of the cricopharyngeal muscle, during thyroidectomy with intraoperative neuromonitoring (IONM).

DETAILED DESCRIPTION:
This study group consisted of a consecutive patients undergoing thyroid surgery with intraoperative neuromonitoring (NIM 3.0 Nerve Monitoring Systeme (Medtronic Xomed, Jacksonville, FL, USA) ) for various diseases. In all patients, each side of the neck operated was considered as a separate entity in our study.

EMG recordings were accomplished with a pair of needle electrodes inserted into the CP and mid-portion of the CT muscle that is located on the superior side of the RLN, which were plugged into the third and fourth channels of interface-connector box, respectively, at the end of the thyroidectomy or lobectomy. The investigators evaluated the innervation pattern of the CT muscle in an other study. Therefore the EBSLN is the main supplier of the CT muscle, the EMG findings of the CT muscle were used to confirm it, in this study.

EBSLN, pharyngeal plexus (PP), RLN and vagus nerve were stimulated with a monopolar stimulator probe at 1 mA. While stimulating these nerves, the ipsilateral CP muscle was visually observed for possible contractions and electromyographic recordings were obtained with the 4-channel NIM 3.0 Nerve Monitoring System.

ELIGIBILITY:
Inclusion Criteria:

* The patients who underwent thyroidectomy.

Exclusion Criteria:

* Preoperative RLN palsy
* Thyroid cancer with massive extrathyroidal extension
* Intentional nerve transection because of cancer invasion
* The assessment failure of nerve function due to the technical deficiency of the IONM equipment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The cricopharyngeal muscle innervation pattern that is evaluated by visual contractions and EMG evoked potentials, with stimulation of the nerves | up to 9 months

SECONDARY OUTCOMES:
The comparison of the EMG amplitudes obtained with the stimulation of the recurrent laryngeal nerve (RLN), vagus nerve, external branch of the superior laryngeal nerve (EBSLN) and pharyngeal plexus. | up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Uludag, Professor, Study Director — Sisli Etfal Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mu L, Sanders I. Neuromuscular specializations within human pharyngeal constrictor muscles. Ann Otol Rhinol Laryngol. 2007 Aug;116(8):604-17. doi: 10.1177/000348940711600809. PMID 17847729
- [Background] Sasaki CT, Kim YH, Sims HS, Czibulka A. Motor innervation of the human cricopharyngeus muscle. Ann Otol Rhinol Laryngol. 1999 Dec;108(12):1132-9. doi: 10.1177/000348949910801207. PMID 10605917
- [Background] Brok HA, Copper MP, Stroeve RJ, Ongerboer de Visser BW, Venker-van Haagen AJ, Schouwenburg PF. Evidence for recurrent laryngeal nerve contribution in motor innervation of the human cricopharyngeal muscle. Laryngoscope. 1999 May;109(5):705-8. doi: 10.1097/00005537-199905000-00005. PMID 10334217
- [Background] Halum SL, Shemirani NL, Merati AL, Jaradeh S, Toohill RJ. Electromyography findings of the cricopharyngeus in association with ipsilateral pharyngeal and laryngeal muscles. Ann Otol Rhinol Laryngol. 2006 Apr;115(4):312-6. doi: 10.1177/000348940611500411. PMID 16676829
- [Result] Oezcelik A, DeMeester SR. General anatomy of the esophagus. Thorac Surg Clin. 2011 May;21(2):289-97, x. doi: 10.1016/j.thorsurg.2011.01.003. PMID 21477778
- [Result] Mu L, Sanders I. The innervation of the human upper esophageal sphincter. Dysphagia. 1996 Fall;11(4):234-8. doi: 10.1007/BF00265207. PMID 8870349
- [Result] Prades JM, Timoshenko AP, Asanau A, Gavid M, Benakki H, Dubois MD, Faye MB, Martin C. [The cricopharyngeal muscle and the laryngeal nerves: contribution to the functional anatomy of swallowing]. Morphologie. 2009 Aug-Sep;93(301):35-41. doi: 10.1016/j.morpho.2009.07.001. Epub 2009 Oct 7. French. PMID 19815444